CLINICAL TRIAL: NCT00291590
Title: Phase 3 Randomized Controlled Trial of the Diabetes Health Enhancement Program for Medicaid and Dual Eligibles in South King County, Washington
Brief Title: Diabetes Health Enhancement Program to Improve Health of People With Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Organization: VA Puget Sound Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: DHEP001
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2006-02-14 (Estimated); Status verified 2005-06

CONDITIONS: Diabetes
Keywords: diabetes; behavioral change; chronic care model; stage of change; Medicaid; Dual eligible; ethnic; self-care
MeSH Terms: conditions — Diabetes Mellitus | interventions — diclofenac hydroxyethylpyrrolidine

INTERVENTIONS:
Behavioral: DHEP

SUMMARY:
Management of chronic diseases, such as diabetes, relies upon the health care providers and the patients self-care. Self management programs for diabetes that target self-empowerment tools have been found to be effective in some studies, but have not typically included individuals on Medicaid.

Our goal for this trial was to observe if patients participating in such a program could decrease glycated hemoglobin levels, improve health status and improve self-care practices.

DETAILED DESCRIPTION:
Design, Setting and Population: A Phase 3, one year prospective trial, randomized to intervention or control (usual care) with Medicaid or dual-Medicare beneficiaries, with diabetes, aged 40-85 years old residing in South King County, Washington.

Intervention: A targeted, multi-component, self-management program incorporating a stage-of-change approach to overcome barriers and facilitate life-style behavior changes to achieve patient-driven health action plans for nutrition or exercise goals.

Main Outcome Measures: Glycemic control (HbA1c), physical and mental health, self-care practices.

Recruitment Status: Completed: participants are no longer being recruited; data analysis is complete.

ELIGIBILITY:
Inclusion Criteria:

* Insured under Medicaid (SSI) or dual enrolled under Medicaid and Medicare for at least one year
* Diagnosed type 1 or type 2 diabetes for at least 1 year (>1 inpatient or >2 outpatients visits with ICD-9 codes 250.00-250.9x, or prescriptions for insulin and/or oral hyperglycemic medications)
* Aged 40-85 years
* Geographically close to the Southeast Senior Center in South King County, Washington, and have a primary care provider (not HMO).

Exclusion Criteria:

* Serious kidney disease (serum creatinine >2.5 or end-stage renal disease)
* Other serious illness that would preclude one-year study participation (dementia, terminal illness, organ transplantation)
* Pregnancy
* Inability to given informed consent.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146
Dates: Start 2001-07; Study Completion 2003-08

PRIMARY OUTCOMES:
Reduction in glycated hemoglobin levels

SECONDARY OUTCOMES:
Improvement in health status and diabetes self-care practices

CONTACTS AND LOCATIONS:
Overall Officials: Gayle E Reiber, PhD, Principal Investigator — Puget Sound VA
Locations (1):
- Puget Sound Veterans Administration, Seattle, Washington, United States

REFERENCES:
- [Background] McFarland LV, Reiber GE, Norman JE. Recruitment of Medicaid and dual-enrolled Medicare beneficiaries with diabetes mellitus into a randomized controlled trial. Am J Manag Care. 2005 Jul;11(7):443-8. PMID 16044981